CLINICAL TRIAL: NCT05188469
Title: A Phase I/IIa (Multi-center, Open-label, Phase I and Multi-center, Open-label, Phase IIa ) Study to Assess the Safety, Tolerability and Explore the Immunogenicity of EG-COVID and EG-COVARo in Healthy Adult Volunteers
Brief Title: Study to Assess the Safety, Tolerability and Explore the Immunogenicity of EG-COVID and EG-COVARo in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EyeGene Inc. (Other)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EG-COVID-102
Record Dates: First submitted 2022-01-06; First posted 2022-01-12 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: COVID-19 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- EG-COVID-003 (Experimental): Subjects will receive one single IM vaccination, the subjects will be enrolled to treatment at a ratio of 1:1 (Phase 1: n=10, Phase 2a: 50 per treatment)
  Component Description (per dose):
  EG-COVID-003 0.5mL (mRNA 100μg)
  Route of administration: Intramuscular injection
  Interventions: Drug: EG-COVID-003
- EG-COVID-001 (Experimental): Subjects will receive one single IM vaccination, the subjects will be enrolled to treatment at a ratio of 1:1 (Phase 1: n=10, Phase 2a: 50 per treatment)
  Component Description (per dose):
  EG-COVID-001 0.5mL (mRNA 200μg)
  Route of administration: Intramuscular injection
  Interventions: Drug: EG-COVID-001
- A: EG-COVID (Experimental): Subjects will receive two single IM vaccinations, 3 weeks apart, the subjects will be enrolled to treatment
  Component Description (per dose):
  EG-COVID 0.5mL (mRNA 400μg)
  Route of administration: Intramuscular injection
  Interventions: Drug: A: EG-COVID
- B: EG-COVID (Experimental): Subjects will receive two single IM vaccinations, 3 weeks apart, the subjects will be enrolled to treatment
  Component Description (per dose):
  EG-COVID 1mL (mRNA 800μg)
  Route of administration: Intramuscular injection
  Interventions: Drug: B: EG-COVID
- C: EG-COVARo (Experimental): Subjects will receive two single IM vaccinations, 3 weeks apart, the subjects will be enrolled to treatment
  Component Description (per dose):
  EG-COVARo 0.5mL (mRNA 800μg)
  Route of administration: Intramuscular injection
  Interventions: Drug: C: EG-COVARo

INTERVENTIONS:
Drug: EG-COVID-003 — Subjects will receive one, two or three single IM vaccination(s), 3 weeks apart, the subjects will be enrolled to treatment at a ratio of 1:1 (Phase 1: n=10, Phase 2a: 50 per treatment)
  EG-COVID-003 0.5mL (mRNA 100μg)
  Route of administration: Intramuscular injection
  Arms: EG-COVID-003
Drug: EG-COVID-001 — Subjects will receive one, two or three single IM vaccinations, 3 weeks apart, the subjects will be enrolled to treatment at a ratio of 1:1 (Phase 1: n=10, Phase 2a: 50 per treatment)
  EG-COVID-001 0.5mL (mRNA 200μg)
  Route of administration: Intramuscular injection
  Arms: EG-COVID-001
Drug: A: EG-COVID — Subjects will receive two single IM vaccinations, 3 weeks apart, the subjects will be enrolled to treatment
  Component Description (per dose):
  EG-COVID 0.5mL (mRNA 400μg)
  Route of administration: Intramuscular injection
  Arms: A: EG-COVID
Drug: B: EG-COVID — Subjects will receive two single IM vaccination(s), 3 weeks apart, the subjects will be enrolled to treatment
  Component Description (per dose):
  EG-COVID 1mL (mRNA 800μg)
  Route of administration: Intramuscular injection
  Arms: B: EG-COVID
Drug: C: EG-COVARo — Subjects will receive two single IM vaccinations, 3 weeks apart, the subjects will be enrolled to treatment
  Component Description (per dose):
  EG-COVARo 0.5mL (mRNA 800μg)
  Route of administration: Intramuscular injection
  Arms: C: EG-COVARo

SUMMARY:
This is Phase 1 and 2a, Multi-center, Open-label study designed to Assess the Safety, Tolerability and Explore the Immunogenicity of EG-COVID and EG-COVARo vaccine in Healthy Adult Volunteers

DETAILED DESCRIPTION:
Subjects will undergo a Screening period beginning up to 14 days prior to enrollment, the vaccination(s) will be administered on Day 0 and Day 21, pre- and post-dose assessment, follow-up visits, and an end of study (EOS) or early termination (ET) visit (as applicable).

Subjects will be enrolled prior to vaccination on Day 0, to one (1) of two (2) or three (3) treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent before the first study-specific procedure;
2. Healthy volunteers aged above 18 years at time of screening;
3. Have received last COVID-19 vaccination more than 3 months ago (more than 90 days) [Only Step 1]
4. Have had at least authorised primary COVID-19 vaccination(s) regardless of numbers of booster. [Only Step 2]
5. The last authorised COVID-19 vaccination, the participants received, should be more than 4 months (16 weeks) prior to the first EG-COVID or EG-COVARo vaccination. [Only Step 2]
6. Participants must have a body mass index (BMI) between ≥18.5 and ≤30.0 kg/m2 at screening;
7. Availability to volunteer for the entire study duration and be willing to adhere to all protocol requirements;
8. Must have a negative urine pregnancy test on the day of dosing prior to each vaccination;
9. Must agree not to donate blood or receive transfusion (including whole blood, plasma, and platelet components).
10. Must agree to use highly effective, medically accepted double-barrier contraception (both male and female partners) from screening until study completion (until 3 months after second vaccination) as specified below in this criterion.

Highly effective double-barrier contraception is defined as use of a condom AND one of the following:

1. Birth control pills (The Pill)
2. Depot or injectable birth control
3. IUD (Intrauterine Device)
4. Birth Control Patch (e.g., Ortho Evra)
5. NuvaRing®
6. Implantable contraception (e.g., Implanon)
7. Documented evidence of surgical sterilisation at least 6 months prior to screening, i.e., tubal ligation for female or vasectomy for male Rhythm methods are not considered as highly effective methods of birth control. Female participants and female partners of male participants must use contraception from the time of informed consent and for 90 days after last vaccination of study drug.

   Female not of childbearing potential must be postmenopausal for ≥12 months. Postmenopausal status will be confirmed through testing of follicle stimulating hormone (FSH) levels ≥ 40 IU/mL at screening for amenorrhoeic female participants.

   Male participants must refrain from sperm donation from start of study and for 90 days after the last vaccination of study drug.

   Female participants who has had hysterectomy at least 6 months prior to screening must provide documented evidence of surgical sterilisation and are not required to use double barrier contraception where this is the usual and preferred lifestyle.

   Participants who are in same-sex relationships are not required to use contraception. Abstinence is acceptable where this is the usual and preferred lifestyle.

   Exclusion Criteria:

   1. Participant with the evidence of COVID-19 infection at screening because of one or more of the following:
   1. Positive for COVID-19 when performing RT-PCR with upper respiratory tract samples; (oropharyngeal/nasopharyngeal swab) (However, if symptoms of cough or sputum are present, additional RT-PCR is performed using a lower respiratory tract sample (sputum), and registration is possible if all are negative)
   2. History of COVID-19 [Step 1 only]; 2. Participant who has the history of COVID-19 infection within 6 months from the first EG-COVID or EG-COVARo vaccination; 3. Close contact with a person infected with COVID-19 within 2 weeks prior to the first EG-COVID or EG-COVARo vaccination; 4. Participants with COVID-19 specific binding antibody titer 1000 IU/mL or less or over 3000 IU/mL (≤ 1000 IU/mL or > 3000 IU/mL) measured by a specific IgG enzyme-linked immunosorbent assay (ELISA) [Step 2 only]; 5. Participant who is considered to have COVID-19 symptoms because of one or more of the following within 2 weeks prior to the first EG-COVID or EG-COVARo vaccination;

   <!-- -->

   1. According to the doctor's opinion, COVID-19 is suspected as a clinical symptom;
   2. History of travel outside of the country and have clinical symptoms of COVID-19; 6. Healthcare workers who can participate in the treatment of COVID-19 patients, or those at high risk of exposure to SARS-CoV-2 (screening clinics and emergency room workers, workers related to COVID-19 prevention, workers involved in collecting or analysing COVID-19 samples, etc.); 7. Clinically significant abnormalities in laboratory tests, electrocardiogram (ECG), or chest X-rays performed at the screening; 8. Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HbsAg), human immunodeficiency virus (HIV) antibody, or Syphilis antibody at Screening; 9. Is acutely febrile or ill 72 hours prior to the first vaccination;

      * Fever is defined as a body temperature ≥38.0°Celsius / ≥100.4°Farenheit.
      * Illness is defined as symptoms due to other infectious diseases (Cough, shortness of breath, chills, muscle pain, headache, sore throat, loss of smell, or loss of taste, etc.) 10. History of a diagnosis or condition that, in the judgment of the Investigator, may affect study endpoint assessment or participant safety, specifically:

   <!-- -->

   1. Respiratory system: asthma, chronic obstructive pulmonary disease (COPD), daily medication administration for active tuberculosis or latent tuberculosis, received treatment due to worsening of respiratory diseases within 5 years prior to the first vaccination
   2. Serious cardiovascular disease: Congestive heart failure, coronary artery disease, myocardial infarction, uncontrolled hypertension, myocarditis, pericarditis, etc.
   3. Nervous system: Epilepsy, seizure (Within 3 years before the first vaccination), migraine, stroke, encephalopathy, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, etc.
   4. Diagnosis of malignancy within the previous 10 years before the first vaccination (except basal cell and squamous cell carcinoma)
   5. Autoimmune diseases, including autoimmune hypothyroidism or psoriasis
   6. Immunodeficiency disease
   7. Hepatobiliary, renal, endocrine, urinary, musculoskeletal or other disorders judged to be clinically significant by the investigator 11. History of SARS-CoV or MERS-CoV infection; 12. History of allergy or hypersensitivity reaction to any components of study vaccine; 13. History of serious adverse reaction, allergy or hypersensitivity reaction to any vaccination; 14. History of platelet-related disease or hemorrhagic disease, or have a history of severe bleeding or bruising after intramuscular injection (IM) or venipuncture, or are taking anticoagulants; (However, according to the judgment of the investigators, there can be involved when using a low dose of an anticoagulant (eg, aspirin at 100mg/day or less)) 15. History of urticaria within 5 years before the first vaccination; 16. History of hereditary or idiopathic angioneurotic edema; 17.History of organ or bone marrow transplantation; 18. History or suspicion of illegal substance use or alcohol abuse within the past 6 months before the first vaccination; 19. Receipt of chronic use of the following drugs within 6 months before the first vaccination:

   <!-- -->

   1. Immunosuppressants and immunomodulators: Azathioprine, cyclosporine, interferon, G-CSF, tacrolimus, everolimus, sirolimus, cyclophosphamide, 6-mercaptopurine, methotrexate, rapamycin, leflunomide, etc.
   2. Systemic steroids: When a dose exceeding 10 mg/day and has been used for more than 14 consecutive days based on prednisolone (However, external steroids, nasal sprays, inhalants, and eye drops are permitted regardless of the dosage) 20. History of dependent psychotropic or opioid drug within 6 months before the first vaccination; 21. Participated in an interventional clinical study except for EG-COVID-102 study (step 1) within 6 months prior to the screening visit or plans to do so while participating in this study; 22. Participant has been vaccinated or plan to vaccinate any within 4 weeks before/after each study vaccine; 23. Participant has received immunoglobulin or blood-derived products within 3 months prior to the first vaccination, or those who plan to administer it during the study; 24. Participant scheduled for surgery while participating in this study; 25. Pregnant or lactating at screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period; 26. Any other reason that, in the opinion of the investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
incidence and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | Day 0 through End of Study (up to 26 weeks after last dose)
  [Safety and Tolerability]
Number of participants with Clinically significant abnormality findings | Day 0 through End of Study (up to 26 weeks after last dose)
  Physical examination finding/s, vital signs, 12-lead electrocardiograms (ECGs), or laboratory test results [Safety and Tolerability]
The incidence and severity of injection site reactions (ISRs) | Day 0 through End of Study (up to 26 weeks after last dose)
  [Safety and Tolerability]

SECONDARY OUTCOMES:
To assess the immune responses profiles of EG-COVID and EG-COVARo in healthy volunteers after vaccinations | Day 0 through End of Study (up to 26 weeks after last dose)
  Participants with a significant increase of anti-SARS-CoV-2 antibodies [Explore the Immunogenicity]

OTHER OUTCOMES:
Ratio of severity of symptoms via COVID-19 infection confirmed by RT-PCR test after 2 weeks of second or third vaccination through end of study (EOS). | Day 0 through End of Study (up to 26 weeks after last dose)
  [Explore the Immunogenicity]

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bloch, A/Prof, Principal Investigator — Holdsworth House
Locations (1):
- Holdsworth House, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No